CLINICAL TRIAL: NCT01750528
Title: The Prevalence and the Progression of Periodontitis in Ankylosing Spondylitis (AS) Patients Versus Non-AS Population
Brief Title: Prevalence and Progression of Periodontitis in Ankylosing Spondylitis
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Yun Jong Lee, Associate Professor, Seoul National University Bundang Hospital
Other Study IDs: IMM 12-0004; IMM 12-0004 (Other Grant/Funding Number: Abbott Labs)
Record Dates: First submitted 2012-09-05; First posted 2012-12-17 (Estimated); Last update posted 2014-06-10 (Estimated); Status verified 2014-06

CONDITIONS: Ankylosing Spondylitis; Periodontitis
MeSH Terms: conditions — Spondylitis, Ankylosing; Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Ankylosing spondylitis: patients aged 18 years or more who meet the 1984 modified New York criteria
- Control: age- (± 3 years) and gender-matched volunteers who do not have inflammatory arthropathy.

SUMMARY:
1. Our hypotheses on the relationship between periodontitis and AS are as follows;

   * The prevalence of periodontitis is higher in AS patients group than that of non-AS control group
   * Anti-TNF-α therapy would favorably affect the disease course of periodontitis.
2. Based on our hypotheses, the specific objectives of the present proposal are as follows;

   * The primary objective is to compare the prevalence rate of periodontitis between AS patient group and non-AS group.
   * The secondary objectives will be:

     * To observe the carriage rate of P. gingivalis in AS and non-AS groups
     * To identify clinical parameters associated with the severity of periodontitis in AS group.
     * To compare the progression of periodontitis at weeks 12 and 24 between AS and non-AS groups or between AS patients with and without anti-TNF-α treatment

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Subjects giving informed written consent
* In case of AS patients, subjects to meet the 1984 modified New York criteria for AS.
* In case of controls, subjects without a history of inflammatory arthropathy

Exclusion Criteria:

* Subjects having received periodontitis treatment including scaling within 6 months before study participation.
* Subjects with a history of taking antibiotics including prophylactic anti-tuberculosis agents within 3 months before study participation.
* Subjects with a hitory of taking immuno-suppresives (methotrexate, leflunomide, tacrolimus, cyclosporin, or azathioprine) or any dose of glucocorticoids (oral or pareneral) within 3 months before study participation.
* Subjects with a history of diabetes mellitus.
* Subjects with aggressive periodontitis requiring open flap debriment at enrollment immediately.
* Subjects with a hitory of clinical inflammatory bowel disease.
* Subjects with active infection, which can make an influence on the levels of acute phase reactants.
* Subjects with any other condition to render the patient unable to understand the scope of the study or preclude the patient from following the protocol in the physician's opinion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. AS group will consist of patients aged 18 years or more who meet the 1984 modified New York criteria for AS.
     i. AS group receiving anti-TNF-α agents will consists of AS patients who have received adalimumab, etanercept, or infliximab before enrollment (or begin anti-TNF-α agents at enrollment) and keep anti-TNF-α agents for 3 months or more after enrollment.
     ii. AS group not receiving anti-TNF-α agents will consists of AS patients who are treated with a non-steroidal anti-inflammatory drug, sulfasalazine, or non-pharmacological therapy and keep non-anti-TNF-α therapy for 3 months or more after enrollment.
  2. Control group will consist of age- (± 3 years) and gender-matched volunteers who do not have inflammatory arthropathy.
Sampling Method: Non-Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2012-09; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
prevalence rate of periodontitis | At enrollment

SECONDARY OUTCOMES:
carriage rate of P. gingivalis | At enrollment
progression of periodontitis | 12 and 24 week

CONTACTS AND LOCATIONS:
Overall Officials: Yun Jong Lee, M.D., Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

REFERENCES:
- [Background] Pischon N, Pischon T, Gulmez E, Kroger J, Purucker P, Kleber BM, Landau H, Jost-Brinkmann PG, Schlattmann P, Zernicke J, Burmester GR, Bernimoulin JP, Buttgereit F, Detert J. Periodontal disease in patients with ankylosing spondylitis. Ann Rheum Dis. 2010 Jan;69(1):34-8. doi: 10.1136/ard.2008.097212. PMID 19126560
- [Derived] Kang EH, Lee JT, Lee HJ, Lee JY, Chang SH, Cho HJ, Choi BY, Ha YJ, Park KU, Song YW, Van Dyke TE, Lee YJ. Chronic Periodontitis Is Associated With Spinal Dysmobility in Patients With Ankylosing Spondylitis. J Periodontol. 2015 Dec;86(12):1303-13. doi: 10.1902/jop.2015.150202. Epub 2015 Aug 20. PMID 26291296